CLINICAL TRIAL: NCT05987969
Title: Efficacy, Tolerability and Safety of a Smartphone-delivered, Fully Automatic Cognitive Behavioural Therapy Programme for Social Anxiety
Brief Title: Efficacy and Safety of the Alena App as a Treatment for Social Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aya Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alena App RCT 2023 #1
Record Dates: First submitted 2023-03-15; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Social Anxiety Disorder (Social Phobia); Social Anxiety; Social Anxiety Disorder
Keywords: RCT; mobile applications; social anxiety; mental health; social anxiety disorder
MeSH Terms: conditions — Phobia, Social; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Access to the "Alena" CBT-based mobile application intervention for 8 weeks. Instructed to complete one of the 4 main modules every 2 weeks. Also asked to complete one additional short exercise per week and engage with one forum post per week.
  Interventions: Other: "Alena" mobile application
- No intervention (No Intervention): Wait list control - Given access to the intervention at the end of the 10-week trial period.

INTERVENTIONS:
Other: "Alena" mobile application — This mobile application primarily comprises CBT-based therapy for social anxiety based on the Clark and Wells model, as well as cognitive assessments, calming exercises and a community forum.
  Arms: Intervention

SUMMARY:
The present study is a randomised controlled trial that seeks to investigate the efficacy and safety of the Alena app as a treatment for social anxiety disorder.

DETAILED DESCRIPTION:
This will be a 10-week web-based parallel-group unblinded randomised controlled trial with an 8-week intervention period and a 2-week follow-up post-intervention. Participants will be randomly allocated to receive access to the Alena app or to a wait list control group, in a 1:1 ratio. The Alena app primarily comprises CBT-based therapy for social anxiety based on the Clark and Wells model, as well as cognitive assessments, calming exercises and a community forum.

ELIGIBILITY:
Inclusion criteria:

* Scored over 30 on the SPIN (indicating at least moderate social anxiety)
* Aged 18 or over
* Fluent in English
* Has access to a smartphone (iOS or Android) and the internet
* UK resident

Exclusion criteria:

* Currently receiving therapy for their mental health
* Mental health medication has changed (dosage or presence) in the last 8 weeks
* Scores over 7 on the AUDIT-C and/or yes on either drug dependence question taken from the DUDIT (indicating drug or alcohol abuse)
* Previous experience with the Alena app through prior studies or user testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Change in Social Phobia Inventory (SPIN) | Change from baseline SPIN at 8 weeks
  The SPIN was designed to assess the full spectrum of symptoms that characterise social anxiety, including fear, avoidance and physiological components.
Change in Work and Social Adjustment Scale (WSAS) | Change from baseline WSAS at 8 weeks
  The WSAS measures the extent to which the respondent's problem impairs their ability to carry out day-to-day activities, such as work, home management and social leisure activities.

SECONDARY OUTCOMES:
Change in Social Phobia Inventory (SPIN) | Change from SPIN level at the end of the intervention period at 4 weeks later
  The SPIN was designed to assess the full spectrum of symptoms that characterise social anxiety, including fear,
Work and Social Adjustment Scale (WSAS) | At the follow-up point of 4 weeks after the end of the intervention period.
  The WSAS measures the extent to which the respondent's problem impairs their ability to carry out day-to-day
Serious adverse events | Within the intervention period of 8 weeks
  Serious adverse events are defined as those that meet the criteria for ISO:14155(A:14)

CONTACTS AND LOCATIONS:
Locations (1):
- Aya Technologies Limited, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garvert MM, McFadyen J, Linke S, McCloud T, Meyer SS, Sobanska S, Sharp PB, Long A, Huys QJM, Ahmadi M. Safety and Efficacy of Modular Digital Psychotherapy for Social Anxiety: Randomized Controlled Trial. J Med Internet Res. 2025 Apr 10;27:e64138. doi: 10.2196/64138. PMID 40208666